CLINICAL TRIAL: NCT05268419
Title: Inhalational Ethanol Therapy (Spray and Nebulized ETHO) in COVID-19 Treatment
Brief Title: Efficacy and Safety of Ethanol Inhalation on COVID-19 Treatment (a Clinical Trial Study)
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ali Amoushahi (Other)
Collaborators: Isfahan University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Ali Amoushahi, Anesthesiology and Critical Care Specialist, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRCT20210725051981N1; U07.1 (Registry Identifier: ICD-10 code); COVID-19, virus identified (Other: ICD-10 code description)
Record Dates: First submitted 2022-02-28; First posted 2022-03-07 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Clinical Infection; Outcome; Morality
Keywords: COVID-19; Ethanol; Inhalation; Nebulizer
MeSH Terms: conditions — Communicable Diseases; COVID-19; Respiratory Aspiration | interventions — Ethanol; Water; Injections

STUDY DESIGN:
Intervention Model Description: Based on the "treatment-on" or "protocol per" strategy, analysis was limited to participants who, according to the study protocol and inclusion criteria, received full interventions and informed the outcomes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding was performed at the level of participants, clinicians, Investigator, nurses and analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethanol inhalation (Active Comparator): 100 ml spray of 35% ethanol were provided and all of participants were instructed to use spray three times every 6 hours from a distance of 20-30 cm from their face, while wearing a mask and closing their eyes, and take a deep breath as they feel nebulized liquid droplets in their nose, mouth, throat, larynx and lungs. Investigators emphasized participants that this protocol must be repeated every six hours to 7 days.
  Interventions: Drug: Ethanol
- Water Distilled inhalation (Placebo Comparator): 100 ml spray of water distilled (placebo) were provided and all of participants were instructed to use spray three times every 6 hours from a distance of 20-30 cm from their face, while wearing a mask and closing their eyes, and take a deep breath as they feel nebulized liquid droplets in their nose, mouth, throat, larynx and lungs. Investigators emphasized participants that this protocol must be repeated every six hours to 7 days.
  Interventions: Drug: Water Distilled

INTERVENTIONS:
Drug: Ethanol — Inhalation of 35%-ethanol spray
  Other Names: Ethyl Alcohol
  Arms: Ethanol inhalation
Drug: Water Distilled — Inhalation of water distilled spray
  Other Names: Water for Injection,Sterile,30Ml
  Arms: Water Distilled inhalation

SUMMARY:
Cytokine storm is the cause of many deaths in COVID -19. The antiviral in-vitro effects of ethanol with solving the fat layer and destroying the glycoprotein of coronavirus have already been established. Proven antiviral effects of ethyl alcohol on extracellular surfaces have been demonstrated by researchers. Immunological studies have shown that acute administration of ethanol can have immunomodulatory effects on innate immunity system mediated by TNFamRNA protein and mitogen-activated protein kinas and reduce cytokine storm by reducing inflammatory factors such as -TLR, TLR, TL-9, interleukin-6 and TL9. It also helps with the chemotaxis of bronchoalveolar macrophages. Other demonstrated effects of ethanol are including: inhibition of virus replication by inhibition of RNA-dependent polymerase, the bronchial dilation by relaxing their involuntary smooth muscles, sedating and relaxation of the participant, muscular analgesic effects.

Ethanol administration has previously been reported for the treatment of methanol poisoning, fat embolism, prevention of preterm labor, pre-eclampsia, and pulmonary edema. The histological safety of inhalation ethanol therapy in the lungs and respiratory tracts of rabbits has been shown by Anna Castro-Balado et al. Ethanol is approved by the Food and Drug Administration. Given these effects of ethanol on virus wall destruction, inhibition of proliferation, and inhibition of immune hyperactivity, the question now is, "Can ethanol inhalation therapy be effective in controlling COVID-19?" There is no a prior knowledge of the inhalation ethanol therapy in COVID-19. This idea was first suggested and published one month after COVID-19 pandemic in Iran (February 2020). To find the answer, a clinical trial was conducted to evaluate the effectiveness of ethanol therapy on clinical state and prognosis of participants. The study was approved by the Medical University of Isfahan, research and ethics committees and is registered at https://irct.ir/trial/58201.

DETAILED DESCRIPTION:
Study Design and Oversight This study is a randomized triple-blind clinical trial with a control group and a parallel design that was conducted at the Isabn-e-Maryam hospital in Medical university of Isfhan, Iran in September 2021. participants randomly assigned in a 1:1 ratio. The study was originally intended for participants admitted to the hospital, but due to amending the country's policy of setting up respiratory clinics in hospitals and prescribing remdesivre and dexamethasone to participants with moderate COVID-19, the study was conducted in this center. Physicians of hospitalized participants were informed about the participant's referral to the respiratory center and this study.

Participants The study population consisted of positive SARS-CoV-2-PCR test. Participants had moderate COVID-19 pneumonia that was referred to the Respiratory Clinic of the Hospital. Inclusion criteria were: agreeing to implement the plan in the form of informed consent, age over 12 years, not pregnant, no history of asthma, alcoholism or epilepsy, no contraindications to ethanol. Exclusion criteria were: intolerance to inhaled ethanol, hypersensitivity or allergies to ethanol, use of drugs that interact with ethanol, and partial or incomplete treatment. Ethanol patch skin test was used to detect possible allergy to alcohol. In this experiment, a drop of ethanol was placed on a gas pad and attached to the participant's arm. After about seven minutes, symptoms such as redness, swelling or itching of the skin will be checked. These symptoms indicated the possibility of allergy or intolerance to alcohol.

Intervention Both control and intervention groups were enrolled with standard treatments based on the national clinical guidelines of Iran. The national standard treatment was intramuscular dexamethasone, 8mg/day (5 days) and 200 mg of remdesivir intravenously on day 1, followed by 100 mg of remdesivir once daily for 4 subsequent days, infused over 30 to 60 minutes. In addition to standard treatment, after obtaining consent, distilled water spray (placebo) was added in the control group and 35% ethanol spray was added in the intervention group. Two sets of 100 ml spray were provided. All of them were instructed to spray three times every 6 hours from a distance of 20-30 cm from their face, while wearing a mask and closing their eyes, and take a deep breath as they feel nebulized liquid droplets in their nose, mouth, throat, larynx and lungs. Investigators emphasized participants that this protocol must be repeated every six hours to 7 days, depending on the persistence of symptoms. How to use it was first taught by investigators and after ensuring the participant's mastery, it was given to the participants to continue at home. In all referrals and follow-ups, the status of spray use was questioned and participants who did not use it or used it irregularly were excluded from the study.

Clinical and Laboratory Monitoring The required information was taken from the participants' records. The data collection sheet had two sections. In the first part were demographic information and underlying diseases. In the second part, clinical information of research cases was written. Data collection checklist was completed by a trained nurse according to clinical symptoms, para-clinical results, clinical examinations and participant's file contents. Data related to research variables including blood oxygen saturation in pulse oximetry, level of inflammatory factor (CRP), need for adjunctive treatment or readmission in hospital and clinical symptoms in both groups were collected until discharge. The Global Symptomatic Score (GSS) was achieved by calculation of cumulative scores of clinical signs and symptoms including fever, headache, body aches, sore throat, runny nose, chills, cough, shortness of breath, anorexia, loss of smell and loss of taste. Any possible side effects were treated in both groups and reported if present. Participants' oxygenation status was monitored and recorded daily with a pulse oximeter. The pulse oximeter was fixed, and at the time of measurement, the participant was breathing room air without receiving supplemental oxygen.

A modified 7-point ordinal scale was used to assess the clinical condition on day 14 of treatment period related to research. This scale has 7 indexes:

1- Death 2. Hospitalized, on invasive mechanical ventilation 3. Hospitalized, on non-invasive ventilation or high flow oxygen devices 4. Hospitalized, requiring low flow supplemental oxygen 5. Hospitalized, for whatever reason, - requiring ongoing medical care (Covid 19 related or otherwise), requiring supplemental oxygen at home.

6. Continue signs or symptoms of Covid 19 without requiring supplemental oxygen - no longer requires ongoing medical care 7. Complete recovery The corrections made to these indicators were due to the limitations that occurred at the same time as the peak of the disease in Iran with the implementation of this study, and participants who needed to be hospitalized were followed up on an outpatient basis in the respiratory clinic. The need for hospitalization in the intensive care unit, drug side effects, clinical symptoms and mortality of the research samples were monitored in two groups. The final follow-up was performed on the 14th day of the disease through telephone calls and review of participants' records and hospital information system documents.

Side effects were recorded after the informed consent was signed and were graded based on version 5.0 of the Common Terminology Criteria for Adverse Event. The required comparisons were performed at 0, 3, 7 and 14 days after the intervention.

Sampling Sampling was performed by an easy random method. Computerized Random number table was used for random assignment. One researcher determined the sequence of random allocations without coordination with other investigators. This person was different from the nurses who assigned participants to the interventions. This person filled the sprays (nebulizer) one by one with 100ml of diluted distilled water or ethanol-35% and labeled them with the numbers coming out of the number container one by one. Investigator assigned a questionnaire and consent form for each spray and wrote the number on the spray in the questionnaire. Each spray was delivered to one of the participants in the study and his / her family or companion was instructed on how to use it. Blinding was performed at the level of participants, clinicians, nurses and analysts.

Statistical Analysis Based on the "treatment-on" or "protocol per" strategy, analysis was limited to participants who, according to the study protocol and inclusion criteria, received full interventions and informed the outcomes. Quantitative and qualitative variables were reported in the form of descriptive statistics including mean standard deviation and number (%), respectively. Quantitative variables with normal and abnormal distributions were compared between groups using independent t-test and Mann-Whitney test, respectively. In addition, qualitative variables were compared between the two groups using Chi-square test.

Comparisons between SPO2 values and clinical symptom scores on days 1, 3, 7 and 14 were performed using a mixed model. Mean changes of baseline values were measured by repeated measures analysis. The sphericity hypothesis was rejected with the help of Mauchly's Statistics and Geisser-Greenhouse correction was used for this purpose.

The proportion of participants who needed additional medical care after 14 days was tested in two groups using χ2 test.

All statistical analyzes were performed using SPSS software version 22 (SPSS Inc., Chicago, IL, USA) and P <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Positive RT-PCR test Less than seven days from onset of symptoms
* Agreeing to implement the plan in the form of informed consent
* Age over 12 years
* Not pregnant
* No history of asthma
* Alcoholism
* Epilepsy
* No contraindications to ethanol

Exclusion Criteria:

* Pregnancy
* Intolerance to inhaled ethanol
* Hypersensitivity
* Allergies to ethanol
* Use of drugs that interact with ethanol
* Partial or incomplete treatment

Ages: 12 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Global Symptomatic Score | day 0
  Global Symptomatic Score (GSS) is considered as an indicator of clinical status of the participants. These included: Fever, Chills, Cough, Headache, Short Breath, Sore throat, Runny nose, Body pain, Anorexia, Anosmia and Lack of taste. Maximum score (6.67) is the worse and minimum score (1.34) mean a better outcome.
Global Symptomatic Score | day 3
  Global Symptomatic Score (GSS) is considered as an indicator of clinical status of the participants. These included: Fever, Chills, Cough, Headache, Short Breath, Sore throat, Runny nose, Body pain, Anorexia, Anosmia and Lack of taste. Maximum score (6.67) is the worse and minimum score (1.34) mean a better outcome.
Global Symptomatic Score | day 7
  Global Symptomatic Score (GSS) is considered as an indicator of clinical status of the participants. These included: Fever, Chills, Cough, Headache, Short Breath, Sore throat, Runny nose, Body pain, Anorexia, Anosmia and Lack of taste. Maximum score (6.67) is the worse and minimum score (1.34) mean a better outcome.
Global Symptomatic Score | day 14th
  Global Symptomatic Score (GSS) is considered as an indicator of clinical status of the participants. These included: Fever, Chills, Cough, Headache, Short Breath, Sore throat, Runny nose, Body pain, Anorexia, Anosmia and Lack of taste. Maximum score (6.67) is the worse and minimum score (1.34) mean a better outcome.

SECONDARY OUTCOMES:
Clinical Status Scale | day 14th
  Clinical status based on the modified 7-point ordinal scale are included:
  1. Death (Lowest scale means the worse outcome)
  2. Hospitalized, on invasive mechanical ventilation
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring low flow supplemental oxygen
  5. Hospitalized, for whatever reason, - requiring ongoing medical care (COVID-19 related or otherwise), requiring supplemental oxygen at home
  6. Continue signs or symptoms of COVID-19 without requiring supplemental oxygen - no longer requires ongoing medical care
  7. Complete recovery (maximum value means the best scale)

OTHER OUTCOMES:
Respiratory status | day 0
  Blood oxygen saturation monitored with pulse oximetry
Respiratory status | day 3
  Blood oxygen saturation monitored with pulse oximetry
Respiratory status | day 7
  Blood oxygen saturation monitored with pulse oximetry
Respiratory status | day 14
  Blood oxygen saturation monitored with pulse oximetry
Inflammatory factor (CRP) | day 0
  WBC counting -CRP titration
Inflammatory factor (CRP) | day 7
  WBC counting -CRP titration
Adverse events | day 0
  Follow-up the participants regarding Ethanol adverse events including: hiccups, eye irritation, cough, shortness of breath, sneezing and unpleasant odor of alcohol.
Adverse events | day 7
  Follow-up the participants regarding Ethanol adverse events including: hiccups, eye irritation, cough, shortness of breath, sneezing and unpleasant odor of alcohol.
Adverse events | day 14
  Follow-up the participants regarding Ethanol adverse events including: hiccups, eye irritation, cough, shortness of breath, sneezing and unpleasant odor of alcohol.
Requires hospitalization | day 7
  Counting the days
Requires hospitalization | day 14
  Counting the days
Requires hospitalization | day 30
  Counting the days
Needing to ICU admission | Day 7
  Evaluate medical file records
Needing to ICU admission | Day 14
  Evaluate medical file records
Needing to ICU admission | Day 30
  Evaluate medical file records
Mortality Rate | Day 7
  Evaluate medical file records
Mortality Rate | Day 14
  Evaluate medical file records
Mortality Rate | Day 30
  Evaluate medical file records

CONTACTS AND LOCATIONS:
Overall Officials: Elham Moazam, Researcher, Study Chair — Chief of Research center of hospital
Locations (1):
- Isabn-e-Maryam Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication are set to be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will become available 6 months after publication.
Access Criteria: It will be available only to researchers working in academic and scientific institutions.
  It is permissible to use this data to find patients who respond better to this treatment.
URL: https://www.researchgate.net/publication/342078305_Elsevier_Editorial_Systemtm_for_Respiratory_Medicine_Manuscript_Draft_Manuscript_Number_Title_A_suggestion_on_Ethanol_therapy_in_COIVDE-19

DOCUMENTS (2):
  • Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT05268419/SAP_000.pdf
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT05268419/ICF_001.pdf